CLINICAL TRIAL: NCT01528007
Title: Treatment of Pathological Gambling With Naltrexone Pharmacotherapy and Brief Intervention - a Placebo Controlled Trial
Brief Title: Treatment of Pathological Gambling With Naltrexone Pharmacotherapy and Brief Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Hannu Alho, Professor, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03062010; 2010-021123-26 (EudraCT Number)
Record Dates: First submitted 2011-10-28; First posted 2012-02-07 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Pathological Gambling
Keywords: Pathological gambling; Treatment intervention
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo pill. (Placebo Comparator)
  Interventions: Drug: Placebo
- 50mg Naltrexone when needed (Active Comparator)
  Interventions: Drug: Naltrexone pharmacotherapy

INTERVENTIONS:
Drug: Naltrexone pharmacotherapy — Naltrexone 50mg when graving to gamble.
  Arms: 50mg Naltrexone when needed
Drug: Placebo — Placebo pill with no active ingredients.
  Arms: Placebo pill.

SUMMARY:
The aim of this research is to explore the efficacy of the opiate antagonist, naltrexone as combined with CBT-intervention in the treatment of pathological gambling (PG). The study period is 2011-2014 during which one hundred Pathological Gamblers will be recruited to participate to this placebo-controlled double-blind trial.

DETAILED DESCRIPTION:
All participants have to be able to read and understand the patient information sheet and sign the informed consent. All participants are free to stop being in the study whenever they wanted. The patients are not paid or reimbursed for participation.

The study periods is 21 weeks during which the participant's have 8 appointments with the researchers. During the meetings research data will be collected and the participant is having Controlled Behavioral Therapy (CBT) consulting from a trained therapist. At the study visits, the subjects are given written instructions for the proper use of naltrexone and advised to take 50 mg naltrexone approximately one hour before gambling or feeling urges to gamble (and to refrain from taking naltrexone at other times). In this study the maximal daily dose is 50mg of naltrexone. The medication is free for the subjects.

ELIGIBILITY:
Inclusion Criteria:

* pathological gambling (scores 5+ from SOGS-R and DSM-IV criteria)

Exclusion Criteria:

* acute hepatitis
* severe liver or kidney dysfunction
* suicide risk or severe depression or other untreated mental health problem
* participation to other gambling research at the same time
* the use of drugs (especially opiates)
* pregnancy
* prisoners
* retarded and mentally ill patients were also excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
PG-YBOCS. | Up to 21 weeks.
  The investigators will interview PG-YBOCS questionnaire from the participants.

SECONDARY OUTCOMES:
Alcohol use. | Up to 21 weeks.
  The investigators will ask the participants to fill in AUDIT questionnaire.
Quality of life. | Up to 21 weeks.
  The investigators will ask the participants to fill in RAND 36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Alho, Professor, Principal Investigator — Finnish Institute for Health and Welfare; Tuuli Lahti, Adjunct Professor, Study Director — Finnish Institute for Health and Welfare
Locations (1):
- National Institute for Health and Welfare, Helsinki, Uusimaa, Finland

REFERENCES:
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734
- [Derived] Kovanen L, Basnet S, Castren S, Pankakoski M, Saarikoski ST, Partonen T, Alho H, Lahti T. A Randomised, Double-Blind, Placebo-Controlled Trial of As-Needed Naltrexone in the Treatment of Pathological Gambling. Eur Addict Res. 2016;22(2):70-9. doi: 10.1159/000435876. Epub 2015 Sep 5. PMID 26339899